CLINICAL TRIAL: NCT05927103
Title: Differences Between Coffee and Non-coffee Drinkers in the Gut Microbiome and Microbiota-Gut-Brain Axis
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Responsible Party: Sponsor
Other Study IDs: APC115a
Record Dates: First submitted 2023-06-02; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Coffee; Microbiome-gut-brain-axis; Stress; Polyphenols; Cognition; Microbiota; Mood; Behaviour; Inflammation
MeSH Terms: conditions — Behavior; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine, stool, blood and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coffee drinkers: Healthy adults between 30 and 50 years-old that consume 3 to 5 cups of caffeinate coffee daily
- Non-coffee drinkers: Healthy adults between 30 and 50 years-old that never consume coffee

SUMMARY:
The aim of this study is to investigate the potential of coffee to act as a prebiotic to alter gut microbiota and improve mood, memory and cognitive performance.

DETAILED DESCRIPTION:
The aim of this study is to investigate the potential of coffee to act as a prebiotic to alter gut microbiota and improve mood, memory and cognitive performance in moderate coffee drinkers compared to non-coffee drinkers healthy adults. Reaction time, socioemotional processing, visual and episodic memory, learning, and an attentional task were administered to measure cognitive performance. Self-report questionnaires on mood, behavior and lifestyle were administered and response to an acute stressor was assessed. Biological samples of saliva, urine, blood, and stool were collected to investigate microbiome-gut-brain-axis signaling such as inflammation, short chain fatty acids and other metabolites production and physiological stress.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Be between 30 and 50 years of age.
3. Be in generally good health as determined by the investigator.
4. Drink moderate amounts of coffee daily (3-5 cups/day)

Exclusion Criteria:

1. Are less than 30 and greater than 50 years of age.
2. Have a significant acute or chronic coexisting illness [cardiovascular, gastrointestinal (GI) [to include functional GI disorders, inflammatory bowel disease, coeliac disease, lactose intolerance, food allergies], immunological, psychiatric [to include formal or as determined by MINI Psychiatric interview, diagnosis of current major depression, anxiety disorder, bipolar spectrum disorder, schizophrenia, other DSM-IV Axis I disorder], neurodevelopmental disorders, immunological, metabolic disorders [to include type I or II diabetes], or any condition which contraindicates, in the investigators judgement, entry to the study,
3. Have a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; all psychoactive medications [to include anxiolytics, antipsychotics, antidepressants, anticonvulsants, centrally acting corticosteroids and opioid pain relievers), laxatives, enemas, antibiotics, anti-coagulants, over-the counter non-steroidal anti-inflammatories (NSAIDS). Subjects should have a wash-out period of 4 weeks.
4. Be hypertensive.
5. Current prebiotic or probiotic supplement use (a wash-out period of 4 weeks after cessation will allow entry to the study), or habitual consumption of foods deemed by the investigator to be particularly rich in prebiotic fibres or probiotic strains or are vegan.
6. Females who are pregnant or planning a pregnancy, or lactating.
7. Participants who are not fluent in English.
8. Participants who have dyslexia or dyscalculia.
9. Are a current habitual daily smoker.
10. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
11. Subjects receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
12. Have a malignant disease or any concomitant end-stage organ disease.
13. Have already done a study in the lab in the past 4 years

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers between 30 and 50 years old.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Gut Microbiota composition | Difference between the groups at baseline.
  Shotgun metagenomics of fecal samples will be performed to quantify the proportion of bacterial taxa within the gut.

SECONDARY OUTCOMES:
Gut microbial metabolites (including Short-Chain fatty acids) | Difference between the groups at baseline.
  Untargeted metabolomics of fecal samples
Coffee-related metabolites | Difference between the groups at baseline.
  Targeted metabolomics of coffee-related metabolomics in fecal and urine samples

OTHER OUTCOMES:
Cognitive performance: attention | Difference between the groups at baseline.
  Assessment of attention using the Paced Auditory Serial Addition Test (PASAT)
Cognitive performance - Episodic memory | Difference between the groups at baseline.
  Assessment of episodic memory using the Modified Rey Auditory Verbal Learning Test (ModRey)
Cognitive performance - Learning and visual memory | Difference between the groups at baseline.
  Assessment of learning and visual memory using the Paired Associates Learning task
Cognitive performance - Processing speed | Difference between the groups at baseline.
  Assessment of processing speed using the Motor Screening Test
Cognitive performance - socioemotional processing | Difference between the groups at baseline.
  Assessment of socioemotional processing using the Emotion Recognition Task
Responses to acute stressor | Difference between the groups at baseline.
  Self-report mood and cortisol responses to the Socially Evaluated Cold Pressor Test
Inflammatory profile | Difference between the groups at baseline.
  Inflammatory markers analysis in LPS-stimulated blood and in the plasma using MSD multiplex technology. The inflammatory markers analyzed were: C-reactive protein, IL6,IL10,IL8, INFgamma, TNFalpha, IL1beta
Cortisol awakening response | Difference between the groups at baseline.
  Cortisol awakening response measurement using ELISAs
Self-reported questionnaires | Difference between the groups at baseline.
  Completion of self-reported questionnaires on mood, depression, anxiety, impulsivity, emotional reactivity, stress, and sleep quality. Low scores represents better outcomes.
Genotyping adenosine receptor A2A | Difference between the groups at baseline.
  Genotyping of 2 SNPs (specifically rs5575187 and rs2298383) of the A2A receptor (ADORA2A) from blood using I-PLEX golden chemistry, Mass array, Mass spectrometry system.

CONTACTS AND LOCATIONS:
Overall Officials: John F Cryan, PhD, Principal Investigator — UCC
Locations (1):
- University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No